CLINICAL TRIAL: NCT03714308
Title: Intravitreal Aflibercept in Neovascular Age-related Macular Degeneration (nAMD): an Observational Study Assessing Patient Relevant Outcomes, Real-world Treatment Pattern and Effectiveness
Brief Title: Aflibercept Injection Into the Vitreous Body of the Eye: Study to Learn More About Patient Relevant Outcomes, Real World Treatment Patterns and How Well the Treatment Works for Patients Suffering From Abnormal Growth of New Blood Vessels Under the Retina.
Acronym: ANDROMEDA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19756
Record Dates: First submitted 2018-09-25; First posted 2018-10-22 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Macular Degeneration
Keywords: Neovascular age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with nAMD_Treatment-naive (anti-VEGF naive): Observational period of therapy with intravitreal aflibercept (IVT-AFL) up to a maximum of 24 months
  Interventions: Drug: Ivt. Aflibercept (Eylea, BAY86-5321)
- Patients with nAMD_Pre-treated with IVT-AFL: Observational period of therapy with intravitreal aflibercept (IVT-AFL) up to a maximum of 24 months
  Interventions: Drug: Ivt. Aflibercept (Eylea, BAY86-5321)
- Patients with nAMD_Pre-treated with any anti-VEGF: Observational period of therapy with intravitreal aflibercept (IVT-AFL) up to a maximum of 24 months
  Interventions: Drug: Ivt. Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Ivt. Aflibercept (Eylea, BAY86-5321) — Treatment is applied according to routine clinical practice and independent of the study setting.

SUMMARY:
In this clinical study researchers want to gain a deeper understanding of treatment consistence under real world conditions over the course of 24 months of Aflibercept injections into the eye for patients suffering from abnormal growth of new blood vessels under the retina (neovascular age-related macular degeneration). The study aims to identify potential reasons that may allow classification of non-consistence as patient or physician driven. They want to describe treatment effectiveness (how well the treatment works) and associations between treatment effectiveness, non-consistence and patient relevant outcomes, such as vision specific quality of life and treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neovascular age-related macular degeneration
* Decision to initiate treatment with intravitreal aflibercept was made as per investigator's routine treatment practice or current treatment with IVT-AFL (all prior anti-VEGF treatments must have been applied by the participating study site)
* No participation in an investigational program with interventions outside of routine clinical practice
* No contra-indications according to the local marketing authorization/ Summary of Product Characteristics (SmPC)
* Ability and willingness to participate in telephone interviews

Exclusion Criteria:

* Any prior therapy with intravitreal steroids in the study eye.
* Concomitant therapy (except nutritional supplements) with any other agent to treat nAMD in the study eye
* Any prior transpupillary thermotherapy, photodynamic therapy, macular rotation/ translocation or macular laser in the study eye or
* Structural damage to the center of the macula in either eye
* Any other condition expected to permanently limit visual acuity outcomes over the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neovascular age-related macular degeneration (nAMD)
Sampling Method: Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Time to first appearance of non-consistence | Up to 24 months
  Non-consistence is:
  * Failure of subjects to appear to a scheduled injection visit;
  * Strong time deviation of injections from approved aflibercept posology.
Reasons why a patient failed to appear to a scheduled injection visit | Up to 24 months
  Asked in telephone interviews

SECONDARY OUTCOMES:
Change in best corrected visual acuity (BCVA) letters | From baseline to 4, 12 and 24 months
Change in central retinal thickness (CRT) | From baseline to 4, 12 and 24 months
Treatment satisfaction by MAC-TSQ | At 4, 12 and 24 months
  Treatment satisfaction is assessed with the MAC-TSQ (Macular Disease Treatment Satisfaction Questionnaire) consisting of 14 items (each item is scored from 0-6) resulting in a score range of 0-72 (a higher score represents better treatment satisfaction).
Change in treatment satisfaction | From 4 month to 12 and 24 months
  Comprises change in treatment satisfaction from 4 months to 12 and 24 months. Treatment satisfaction is assessed with the MAC-TSQ (Macular Disease Treatment Satisfaction Questionnaire) consisting of 14 items (each item is scored from 0-6) resulting in a score range of 0-72 (a higher score represents better treatment satisfaction).
Vision-specific quality of life by NEI VFQ-25 | At baseline, 4, 12 and 24 months
  Vision-specific quality of life is assessed with the NEI VFQ-25 (National Eye Institute Visual Function Questionnaire), i.e. a 25-item questionaire that gives a score on a scale from 0 (worst) to 100 (best = no vision problems).
Change in vision-specific quality of life | From baseline to 4, 12 and 24 months
  Comprises change in vision-specific quality of life between baseline and 4, 12 and 24 months. Vision-specific quality of life is assessed with the NEI VFQ-25 (National Eye Institute Visual Function Questionnaire), i.e. a 25-item questionaire that gives a score on a scale from 0 (worst) to 100 (best = no vision problems).
Burden of therapy | At 4, 12 and 24 months
  Descriptive measure summarising information about patient´s time for scheduling and attending appointments and anxiety reasons. Asked in telephone interviews.
Information about disease and treatment | At 4, 12 and 24 months
  Describes to what extent patients were informed about their disease and treatment. Asked in telephone interviews.
Willingness to continue therapy | At 4, 12 and 24 months
  Asked in telephone interviews
Reasons for treatment discontinuation | At 4, 12 and 24 months
  Asked in telephone interviews
Change in general quality of life by EQ-5D | From baseline to 12 and 24 months
  General quality of life is assessed with EQ-5D ®, a 5-item questionnaire assessing 5 health related dimensions on 5 levels (% is calculated for each level) and complemented by a visual analogue scale (range 0-100, high score represents better quality of life).
Percentage of non-persistent patients | At 12 and 24 months
  Non-persistence is:
  Patients terminating treatment with aflibercept.
Time from baseline to first instance of non-persistence | Up to 24 months
  Non-persistence:
  Patients terminating treatment with aflibercept.
Percentage of patients receiving 3 initial monthly injections | Up to 24 months
Percentage of consistently treated patients | At 12 and 24 months
  Non-consistence is:
  * Failure of subjects to appear to a scheduled injection visit;
  * Strong time deviation of injections from approved aflibercept posology.
Proportion of patients undergoing therapeutic switch | At 12 and 24 months
Reasons for therapeutic switching | At 12 and 24 months
  Asked in telephone interviews
Proportion of patients discontinuing disease monitoring at participating center | At 12 and 24 months
Average time between visits | Up to 24 months
Average time between injections in the study eye | Up to 24 months
Number of injections in the study eye per year | Up to 24 months
Number of visits per study eye per year | Up to 24 months
  Comprises monitoring, injection and post-injection visits
Number of visits in clinics/ ophthalmology practices other than the study center per year | Up to 24 months
Number of examinations of the study eye per year | Up to 24 months
  Comprises optical coherence tomography (OCT), visual acuity tests, funduscopy examinations or angiography examinations.
Number of injections until start of observation | At baseline
  Only for pre-treated patients
Duration of treatment until start of observation | At baseline
  Only for pre-treated patients
Type of treatment until start of observation | At baseline
  Only for pre-treated patients

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.